CLINICAL TRIAL: NCT05609084
Title: Intensive Preoperative Speech Rehabilitation in Drug-Resistant Temporal Epilepsy
Acronym: REPREO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-17; ID-RCB (Other: 2021 - A03232-39)
Record Dates: First submitted 2022-10-25; First posted 2022-11-08 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy; Anomia; Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy; Anomia; Epilepsy, Temporal Lobe | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Other): Patients will have speech therapy assessment in addition to standard care.
  Interventions: Procedure: Speech therapy assessment
- Experimental (Experimental): Patients will have speech therapy assessment and intensive speech rehabilitation
  Interventions: Procedure: Speech therapy; Procedure: Speech therapy assessment

INTERVENTIONS:
Procedure: Speech therapy — Patients will connect on an interface to pratice speech therapy
  Arms: Experimental
Procedure: Speech therapy assessment — Patients will be followed by an speech therapist

SUMMARY:
Out of 30,000 new cases per year in France, 30% of epileptic patients are drug-resistant. Neurosurgery, which consists in resecting the epileptogenic zone, is the only chance of cure. In the case of temporal epilepsy of the language-dominant hemisphere (TLE), this procedure presents a high risk of increasing cognitive difficulties and may even be contraindicated for this reason alone. The difficulties found are impairments in lexical access (anomia) and verbal memory and affect more than 60% of patients . Preoperative cognitive rehabilitation could influence brain plasticity mechanisms but there are currently no recommendations on this topic. In this context, the investigators have developed a speech rehabilitation procedure specific to the needs of ELTPR patients. They rely on cognitive hypotheses explaining the disorders but also on models of rehabilitation-induced neural plasticity likely to improve cognitive reserve before surgery. The investigators hypothesize that preoperative cognitive language rehabilitation in ELTPR patients may decrease surgical risk and improve postoperative language prognosis.

The primary objective is to demonstrate the protective efficacy of preoperative speech rehabilitation on language performance postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 16 years of age and older,
2. Patient whose epileptogenic area involves the temporal structures of the hemisphere specialized for language,
3. Patient whose hemispheric specialization for language is known
4. Patient willing to undergo resective surgery such as anterior temporal lobectomy or resection in the temporal lobe involving the hippocampus and/or the baso-temporal language area and whose planned surgery date is compatible with the performance of the study,
5. Patient with a known NTB score
6. Patient who has signed an informed consent or patient whose parents or legal guardians have signed the informed consent (or a single parent or legal guardian if applicable)
7. Patient whose first language is French (1st language learned by the patient),
8. Patient declaring to be familiar with the use of a computer and having access to an internet connection from home
9. Patient affiliated or benefiting from a social security system.

Exclusion Criteria:

1. Patient with a speech disorder that may impair intelligibility and compromise the use of the interface;
2. Patient with an uncorrected hearing impairment,
3. Patients with a total intelligence quotient (IQ) <70 (assessed in the context of care, in the year preceding the surgical procedure)
4. Patients who are pregnant, nursing, deprived of liberty, under guardianship or curatorship.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Effect of rehabilitation on immediate postoperative performances | Day 7 after surgery
  Number of images quoted

SECONDARY OUTCOMES:
Impact of rehabilitation on long-term postoperative performance | 6 months after surgery
  Number of images quoted
Impact of rehabilitation on immediate on standardized language tests | Day 7 after surgery
  % of correct answers of language tests
Impact of rehabilitation on long-term postoperative performance on standardized language tests | 6 months after surgery
  % of correct answers of language tests
Impact of preoperative rehabilitation on verbal memory | Day 7 after surgery
  Verbal memory task
Impact of preoperative rehabilitation on verbal memory | 6 months after surgery
  Verbal memory task
Lexical fluency | Day 7 after surgery
  Lexical evocation tests limited to 2 minutes according to a formal criterion or an imposed categorical criterion
Lexical fluency | 6 months after surgery
  lexical evocation tests limited to 2 minutes according to a formal criterion or an imposed categorical criterion
Denomination of control lists | Day 7 after surgery
  Number of words quoted
Denomination of control lists | 6 months after surgery
  Number of words quoted
Self-reported perception of anomia | Day 7 after surgery
  Use of an ad-hoc scale graduated from 0 (no complaint) to 10 (maximum complaint)
Self-reported perception of anomia | 6 months after surgery
  Ad-hoc scale graduated from 0 (no complaint) to 10 (maximum complaint)
Evaluation of Quality of life | Day 7 after surgery
  Quality Of Life in Epilepsy Inventory (QOLIE-31) (0 meaning better outcome, highest score meaning worse outcome)
Evaluation of Quality of life | 6 months after surgery
  Quality Of Life in Epilepsy Inventory (QOLIE-31) (0 meaning better outcome, highest score meaning worse outcome)
Impact of pre-operative rehabilitation on the number of post-operative rehabilitation sessions | 6 months after surgery
  Number of speech therapy sessions performed postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Francois CREMIEUX, Study Director — AP-HM
Locations (12):
- France (12):
  - Service EFSN - Hôpital Pellegrin, Bordeaux
  - Service de Neurologie de l'Epilepsie - CHU Grenoble-Alpes, Grenoble
  - Département de Neurophysiologie Clinique - Hôpital Roger Salengro - CHU Lille, Lille
  - Hôpital Neurologique Pierre Wertheimer- Service de Neurologie Fonctionnelle et Epileptologie - Hospices Civils Lyon, Lyon
  - Service Epilptologie et Rythmologie Cérébrale, Marseille
  - Service de Neurologie - Hôpital central -CHU Nancy, Nancy
  - Département de Neurologie - Hôpital de la Pitié-Salpêtrière - APHP, Paris
  - Service de Neurochirurgie -GHU Sainte-Anne, Paris
  - Service de Neurologie - Fondation ophtalmologique de Rothschild - Fondation Rothschild, Paris
  - Service de Neurologie - CHU de Rennes, Rennes
  - Service de Neurologie - Hôpitaux Universitaires, Hôpital de Hautepierre, Strasbourg
  - Explorations Neurophysiologiques, Pôle des Neurosciences - Hôpital Pierre Paul Riquet, Purpan, Toulouse